CLINICAL TRIAL: NCT05002816
Title: Novel Combination of Belantamab Mafodotin and Elotuzumab to Enhance Therapeutic Efficacy in Multiple Myeloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Natalia Neparidze, Assistant Professor, Medical Oncology, Hematology & Oncology, Yale University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000028918
Record Dates: First submitted 2021-07-21; First posted 2021-08-12 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-09

CONDITIONS: Multiple Myeloma
Keywords: Belantamab Mafodotin; Elotuzumab
MeSH Terms: conditions — Multiple Myeloma | interventions — elotuzumab; belantamab mafodotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Belantamab Mafodotin and Elotuzumab Arm (Experimental): Elotuzumab will be administered via intravenous infusion at an established dose of 10 mg/kg on days 1, 8, 15, 22 every 28 days for cycles 1 and 2, followed by 20mg/kg on day 1 of each cycle thereafter, cycles repeated every 28 days.
  Belantamab mafodotin will be administered via IV infusion. There will be 3 dose levels for belantamab mafodotin, with the starting dose of 1.9 mg/kg IV at every 4 week interval. Up to 12 subjects will be treated at this dose level. If the initial dose is found to be too toxic, dose of belantamab mafodotin 1.9 mg/kg every 8 weeks will be tested, further dose reduction to 1.4mg/kg every 8 weeks will be administered.
  Interventions: Drug: Elotuzumab; Drug: Belantamab mafodotin

INTERVENTIONS:
Drug: Elotuzumab — Elotuzumab will be administered via intravenous infusion at an established dose of 10 mg/kg on days 1, 8, 15, 22 every 28 days for cycles 1 and 2, followed by 20mg/kg on day 1 of each cycle thereafter, cycles repeated every 28 days.
Drug: Belantamab mafodotin — Belantamab mafodotin will be administered via IV infusion on day 1 of each 28 day cycle. There will be 3 dose levels for belantamab mafodotin, with the starting dose of 1.9 mg/kg IV at every 4 week interval. Up to 12 subjects will be treated at this dose level. If the initial dose is found to be too toxic, dose of belantamab mafodotin 1.9 mg/kg every 8 weeks will be tested, further dose reduction to 1.4mg/kg every 8 weeks will be administered. Following the dose evaluation, there will be a dose expansion cohort wtih 12 additional subjects. There is no dose escalation planned in this study.

SUMMARY:
The purpose of this research study is to determine if two drugs approved for treating multiple myeloma, belantamab mafodotin and elotuzumab, are safe and more effective when used together.

DETAILED DESCRIPTION:
Patients with RR MM beyond two-three lines of therapy have inferior outcomes. They have to cycle through the available lines of treatment options and ultimately succumb to progressive disease. Despite improvements in modern treatments this subset of MM patients has a grim prognosis and thus represent a population with unmet need. Hence, further advances in combination therapies are required. MM is associated with both qualitative and quantitative T cell dysfunction owing to variety of mechanisms including increased expression of inhibitory immune checkpoint molecules. Elotuzumab enhances NK cell cytotoxicity via SLAMF7 ligation and has an established role in therapy of RR MM in combination with immunomodulatory agents (iMIDs). On the other hand, BCMA has emerged as one of the best therapeutic targets to eradicate plasma cells in MM. Therapeutic success with anti-BCMA ADC belantamab mafodotin is readily evident based on the results of recent trials DREAMM 1 and DREAMM2 in relapsed/refractory MM, leading to its Breakthrough Therapy Designation awarded by US FDA in 2017. Bela has demonstrated the potential to induce immunogenic cell death (ICD) in a BCMA-expressing MM cells. Tumor cells undergoing ICD induced an antigen-specific T cell response, enhancing anti-tumor effects. Generally, in myeloma, success in therapy has always been achieved by multifaceted treatment approach, targeting several pathways concurrently. To combat antigen loss and resistance, combining monoclonal antibodies with different targets is proposed. In this study, we propose immune-stimulatory therapy with anti-SLAMF7 antibody elotuzumab in combination with belantamab mafodotin in subjects with RR MM. Administration of elotuzumab would enrich NK cells and together with belantamab mafodotin would further intensify anti-tumor immunity against MM. This combination would provide a novel all-immune targeted therapy with potentially increased efficacy.

The investigators expect that this unique combination of an antibody drug conjugate and an immune-stimulatory monoclonal antibody, targeting two very relevant pathways in MM will result in significant clinical benefit for patients with RR MM. From the standpoint of safety, each one of these immune-pharmaceutical drugs separately is well-tolerated, and in combination are not expected to display overlapping toxicity. Thus, the investigators believe, the adverse event profile of this combination would be favorable.

The phase I portion of the study was completed successfully. Phase II portion of the study is actively enrolling.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must have MM that has relapsed after or is refractory to at least 3 prior lines of therapy. Relapsed/refractory disease as defined by IMWG criteria.
2. Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
3. Participant must be ≥ 18 years of age
4. Prior line of therapy must include iMID, proteasome inhibitor, and anti-CD38 monoclonal antibody. Prior elotuzumab is allowed.
5. Participant must have adequate organ function, defined as:

   * ANC ≥0.5X 10 9/L
   * Hemoglobin ≥8.0 g/dL
   * Platelets ≥50X 10 9/L
   * Total bilirubin ≤1.5X ULN (Isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%)
   * ALT ≤2.5 X ULN
   * eGRF ≥30 mL/min/ 1.73 m2
   * Spot urine (albumin/creatinine ratios) <500 mg/g (56 mg/mmol) OR
   * Urine dipstick Negative/trace (if ≥1+ only eligible if confirmed <500 mg/g (56 mg/mmol) by albumin/creatinine ratio (spot urine from first void)
6. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies::
   * Is not a woman of childbearing potential (WOCBP) OR
   * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), preferably with low user dependency (as described in Appendix 3), during the intervention period and for at least 4 months after the last dose of study intervention and agrees not to donate eggs (ova, oocytes) for the purpose of reproduction during this period. The investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study intervention.

   A WOCBP must have a negative highly sensitive serum pregnancy test (as required by local regulations) within 72 hours before the first dose of study intervention.

   The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.

   Nonchildbearing potential is defined as follows (by other than medical reasons):
   * ≥45 years of age and has not had menses for >1 year
   * Patients who have been amenorrhoeic for <2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
   * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.
7. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies.

   Male participants are eligible to participate if they agree to the following during the intervention period and for 6 months after the last dose of study treatment to allow for clearance of any altered sperm:

   • Refrain from donating sperm

   PLUS either:

   • Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent.

   OR

   • Must agree to use contraception/barrier as detailed below: Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females)
8. All prior treatment-related toxicities (defined by National Cancer Institute- Common Toxicity Criteria for Adverse Events (NCI-CTCAE), version 5.0) must be ≤ Grade 2 at the time of enrolment except for alopecia.
9. Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent

Exclusion Criteria:

1. Participant must not have current corneal epithelial disease except mild changes in corneal epithelium
2. Participant must not have current unstable liver or biliary disease defined by the presence of ascites, encephalopathy, esophageal or gastric varices, persistent jaundice, or cirrhosis. Note: Stable non-cirrhotic chronic liver disease (including Gilbert's syndrome or asymptomatic gallstones) or hepatobiliary involvement of malignancy is acceptable if otherwise meets entry criteria
3. Participant must not have presence of active renal condition (infection, requirement for dialysis or any other condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM and stable chronic kidney disease are eligible, provided they fulfil inclusion criteria
4. Participant must not use contact lenses while participating in this study
5. Participant must not be simultaneously enrolled in any other interventional clinical trial
6. Participant must not have used an investigational drug or approved systemic anti- myeloma therapy (systemic steroids are allowed) within 14 days preceding the first dose of study drug
7. Participant must not have had plasmapheresis within 7 days prior to first dose of study treatment
8. Participant must not have received prior treatment with a monoclonal antibody within 30 days of receiving the first dose of study drugs
9. Participant must not have had major surgery ≤ 4 weeks prior to initiating study treatment
10. Participant must not have any evidence of active mucosal or internal bleeding
11. Participant must not have evidence of cardiovascular risk including any of the following:

    * Evidence of current clinically significant uncontrolled arrhythmias, including clinically significant ECG abnormalities such as 2nd degree (Mobitz Type II) or 3rd degree atrioventricular (AV) block.
    * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within three (3) months of Screening.
    * Class III or IV heart failure as defined by the New York Heart Association functional classification system [NYHA, 1994]
    * Uncontrolled hypertension
12. Participant must not have known immediate or delayed hypersensitivity reaction or idiosyncratic reactions to belantamab mafodotin or drugs chemically related to belantamab mafodotin, or any of the components of the study treatment
13. Participant must not have an active infection requiring IV antimicrobial treatment
14. Participant must not have known HIV infection
15. Participant must not have presence of hepatitis B surface antigen (HBsAg), or hepatitis B core antibody (HBcAb) at screening or within 3 months prior to first dose of study treatment
16. Participant must not have positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months prior to first dose of study treatment.

    Note: Participants with positive Hepatitis C antibody due to prior resolved disease can be enrolled, only if a confirmatory negative Hepatitis C RNA test is obtained.

    Note: Hepatitis RNA testing is optional and participants with negative Hepatitis C antibody test are not required to also undergo Hepatitis C RNA testing.
17. Participant must not have invasive malignancies other than disease under study, unless the second malignancy has been medically stable for at least 2 years and, in the opinion of the principal investigators, will not affect the evaluation of the effects of clinical trial treatments on the currently targeted malignancy. Participants with curatively treated non- melanoma skin cancer may be enrolled without a 2-year restriction.
18. Participant must not have any serious and/or unstable pre-existing medical, psychiatric disorder, or other conditions (including lab abnormalities) that could interfere with participant's safety, obtaining informed consent or compliance to the study procedures
19. Participants must not be pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2022-02-21 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of elotuzumab in combination with belantamab mafodotin in subjects | 28 days
  Study patients will be enrolled and treated in cohorts of size 4 with maximum of 12 patients in the Phase I portion of the trial with possible dose de-escalation of belantamab mafodotin plus a fixed level of elotuzumab. Starting dose of belantamab mafodotin will be 1.9 mg/kg q4w. If the DLT rate hits de-escalation boundary (≥ 29.8%), four more patients will be enrolled for lower dose level with 1.9 mg/kg q8w; further dose reduction to 1.4mg/kg every 8 weeks will be planned for ongoing toxicity. Otherwise next cohort of 4 will be treated at same dose. The MTD will be determined once the maximum sample size of 12 for phase I portion is reached or stop the trial if 8 patients are treated at the initial dose without need of de-escalation.
Number of Participants who Experienced Dose-Limiting Toxicities (DLTs) | 28 days
  DLT is defined as Grade 3 or greater febrile neutropenia lasting >48 h despite adequate treatment, Grade 4 thrombocytopenia less than 25 accompanied by clinically significant bleeding, any Grade 3 or greater non-hematologic toxicity (other than corneal events) which is more severe than expected for an individual agent or which does not resolve with appropriate supportive treatment within 48 hours, any Grade 3 or greater non-hematologic laboratory value if the abnormality leads to hospitalization, grade 4 Keratopathy Visual Acuity (KVA) Scale, and liver toxicity meeting prespecified liver stopping criteria

SECONDARY OUTCOMES:
Preliminary evaluation of clinical efficacy/response rate | Every 28 day cycle until progression up to 2 years
  Clinical efficacy and response rate will be determined by the MM labs and bone marrow biopsy . The options for overall response rate (ORR) will be: stable disease (SD) partial response (PR), very good partial response (VGPR), complete response (CR) and stringent complete response (sCR) according to the 2016 International Myeloma Working Group (IMWG). Response evaluated with MM labs each cycle and bone marrow biopsy at C3D1.
To evaluate progression free survival (PFS) | Followed for progression free survival until progression up to 2 years
  To evaluate progression free survival (PFS), MM labs (SPEP, serum IFE, serum free light chains/ratio, immunoglobulins, UPEP/IFE) will be conducted every cycle to evaluate disease. Progressive disease will be assessed by standard IMWG response criteria.
To evaluate overall survival (OS) | Followed until loss of follow-up, withdrawal of consent, death from any cause, or termination of study up to 2 years
  To evaluate overall survival (OS), patients will be followed for overall survival under loss of follow-up, withdrawal of consent, death from any cause, or termination of study
To evaluate minimal residual disease (MRD) by multi-parameter flow cytometry and by next-generation sequencing (NGS) | At follow-up visit (30 days +/-3 after discontinuation)
  To evaluate minimal residual disease (MRD) by multi-parameter flow cytometry and by next-generation sequencing (NGS) via bone marrow biopsy at follow-up visit (30 days +/- 3 after discontinuation)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Neparidze, MD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided